CLINICAL TRIAL: NCT03467035
Title: Role of NLRP3 Inflammasone and Hypoxia in the Severity of Osteoporosis in Patients With Bronchiectasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chun-Hua Wang, MD (Other)
Responsible Party: Sponsor-Investigator, Chun-Hua Wang, MD, professor, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Other Study IDs: 201701317A3
Record Dates: First submitted 2018-03-07; First posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Bronchiectasis Adult; Osteoporosis, Osteopenia
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — The remaining samples after the completion of this study are deposited in the Human Genome Database of Chang Gung Memorial Medical Center _ Linkou __ Chang Gung Memorial Hospital for the follow-up study (including gene research) approved by the Human Ethics Committee of the Hospital
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- desaturation: ΔSpO2 >10% or lowest SpO2<90 during baseline six minute walk test
  Check serum level of inflammasone, such as IL-1beta, TGF-beta TRT-PCR for PBMC
  Interventions: Other: Inflammasone
- non-desaturation: ΔSpO2 <10% and lowest SpO2>90 during baseline six minute walk test
  Check serum level of inflammasone, such as IL-1beta, TGF-beta TRT-PCR for PBMC
  Interventions: Other: Inflammasone

INTERVENTIONS:
Other: Inflammasone — Serum level of cytokine and RT-PCR for PBMC

SUMMARY:
The objectives of this research grant are to determine the association of hypoxia with the severity of osteoporosis in the patients with bronchiectasis and whether the mechanism of inflammation is triggered by inflammasones, which makes it more prone to osteoporosis in patients with bronchiectasis.

DETAILED DESCRIPTION:
80 patients with proven bronchiectasis, diagnosed by high-resolution computed tomography (HRCT), will be recruited from our outpatient clinic of Chang Gung Memorial Hospital with written informed consent. Inclusion criteria are: daily sputum > 10 ml; absence of asthma or other unstable systemic diseases; and "steady-state" bronchiectasis (< 10% alteration of 24 h sputum volume, FEV1, and FVC, and in the absence of deterioration in respiratory symptoms at baseline visits). Exclusion criteria include: unreliable clinic attendance; regular user of inhaled or oral corticosteroids; history of lung resection and known asthma defined according to American Thoracic Society guidelines.

The lung function and desaturation will be assessed by six-minute walking tests and the severity of disease will be evaluated by HRCT scores. Peripheral blood sample (40ml/person) is performed to analyze the bone turnover markers and the level of Hif in PBMC.

ELIGIBILITY:
Inclusion Criteria:

1. willing to sign a written consent form
2. Male and female subjects with bronchiectasis diagnosed by high-resolution computed tomography
3. willing to accept 6-minute exercise pulmonary function test and blood draw
4. Men and women over the age of 20
5. Has undergone chest computed tomography and bone density examination in the recent five years

Exclusion Criteria:

1. pregnant women or lactating women
2. asthma, lung resection history before the screening period
3. active Tuberculosis infection
4. Have received oral steroid treatment within 30 days
5. current acute attack or clinical symptoms instability of bronchiectasis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 adult patients with proven bronchiectasis, diagnosed by high-resolution computed tomography (HRCT), will be recruited from our outpatient clinic of Chang Gung Memorial Hospital with written informed consent. The inclusion and exclusion criteria are described above.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-12-21 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
six minute walk test | 6 months
  six minute walk test distance

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Hua Wang, Study Director — Chang Chung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cole PJ. Inflammation: a two-edged sword--the model of bronchiectasis. Eur J Respir Dis Suppl. 1986;147:6-15. PMID 3533593
- [Background] Arnett TR. Acidosis, hypoxia and bone. Arch Biochem Biophys. 2010 Nov 1;503(1):103-9. doi: 10.1016/j.abb.2010.07.021. Epub 2010 Jul 23. PMID 20655868
- [Background] Utting JC, Flanagan AM, Brandao-Burch A, Orriss IR, Arnett TR. Hypoxia stimulates osteoclast formation from human peripheral blood. Cell Biochem Funct. 2010 Jul;28(5):374-80. doi: 10.1002/cbf.1660. PMID 20556743
- [Background] Kim RY, Pinkerton JW, Gibson PG, Cooper MA, Horvat JC, Hansbro PM. Inflammasomes in COPD and neutrophilic asthma. Thorax. 2015 Dec;70(12):1199-201. doi: 10.1136/thoraxjnl-2014-206736. Epub 2015 Oct 22. No abstract available. PMID 26493990
- [Background] Diehl N, Johnson MM. Prevalence of Osteopenia and Osteoporosis in Patients with Noncystic Fibrosis Bronchiectasis. South Med J. 2016 Dec;109(12):779-783. doi: 10.14423/SMJ.0000000000000565. PMID 27911973
- [Background] McDonnell MJ, Aliberti S, Goeminne PC, Restrepo MI, Finch S, Pesci A, Dupont LJ, Fardon TC, Wilson R, Loebinger MR, Skrbic D, Obradovic D, De Soyza A, Ward C, Laffey JG, Rutherford RM, Chalmers JD. Comorbidities and the risk of mortality in patients with bronchiectasis: an international multicentre cohort study. Lancet Respir Med. 2016 Dec;4(12):969-979. doi: 10.1016/S2213-2600(16)30320-4. Epub 2016 Nov 16. PMID 27864036